CLINICAL TRIAL: NCT05049954
Title: The Effect of a Healthy Ketogenic Diet Versus Calorie-restricted Low Fat Diet on Weight Loss and Metabolic Outcomes for Obesity: A Randomised Controlled Trial
Brief Title: Weight Loss for a Healthier You Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/00833
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2021-09

CONDITIONS: Ketogenic Dieting; Weight Loss; Obesity; Metabolic Syndrome
Keywords: Low carbohydrates; mHealth; Randomized controlled trial
MeSH Terms: conditions — Weight Loss; Obesity; Metabolic Syndrome | interventions — Diet, Reducing

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, participants in the HKD group will be advised to follow a calorie-restricted healthy ketogenic diet (n=35), with a maximum of 50g net carbohydrate intake daily. Those in the control group will be instructed to follow a calorie-restricted low fat diet (LFD) (n=35).
Masking Description: It is not feasible to apply blinding to the study design due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Ketogenic Diet (HKD) (Experimental): Participants in the HKD group will be advised to follow a calorie-restricted healthy ketogenic diet (n=35), with a maximum of 50g net carbohydrate intake daily, with calorie prescriptions calculated based on the Schofield equation, adjusted with a deficit of 500 kcal daily to promote weight loss.
  Participants will attend group workshops conducted by dietitians at weeks 1, 3, 5, 7, and thereafter at 6-week intervals over the course of a 6-month period (total of 7 workshops). Participants will also be recommended to use the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, steps count and to aid in their adherence to the diet and physical activity recommendations during the 6 months period. The participants will be recommended to achieve their incremental daily step count goal from 3,000, 7,000 to 10,000 to promote increased physical activity, as per their tolerance.
  Interventions: Other: Calorie-Restricted Healthy Ketogenic Diet
- Low Fat caloric-restricted Diet (LFD) (Active Comparator): Participants in the reference group will be instructed to follow a calorie-restricted low fat diet (LFD) (n=35), with calorie prescriptions calculated based on the Schofield equation, adjusted with a deficit of 500 kcal daily to promote weight loss.
  Similar to the experimental group, participants will attend group workshops conducted by dietitians at weeks 1, 3, 5, 7, and thereafter at 6-week intervals over the course of a 6-month period (total of 7 workshops). Participants will also be recommended to use the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, steps count and to aid in their adherence to the diet and physical activity recommendations during the 6 months period. The participants will be recommended to achieve their incremental daily step count goal from 3,000, 7,000 to 10,000 to promote increased physical activity, as per their tolerance.
  Interventions: Other: Calorie-Restricted Low Fat Diet

INTERVENTIONS:
Other: Calorie-Restricted Healthy Ketogenic Diet — Participants in the experimental group will be advised on a Calorie-restricted Healthy Ketogenic Diet via 7 workshops. Participants will also be advised to monitor their urinary ketones to track compliance.
  Other Names: Very Low Carbohydrate Diet
  Arms: Healthy Ketogenic Diet (HKD)
Other: Calorie-Restricted Low Fat Diet — Participants will be advised on Calorie-restricted Low Fat diet via 7 workshops.
  Other Names: Weight loss diet
  Arms: Low Fat caloric-restricted Diet (LFD)

SUMMARY:
In view of the research gap in the safety of traditional ketogenic diet, there is a need for a healthy alternative to the ketogenic diet that reduces the individual's propensity to adverse diet choices. Healthy guidelines to be adopted include a diet low in saturated fat, trans fat, and sugar, along with adequate fibre. Potentially with these guidelines in effect, the associated risks for CVD would be reduced. Therefore, this study will investigate the effect of a calorie-restricted healthy ketogenic diet versus a calorie-restricted low fat diet on weight loss and metabolic outcomes among individuals with obesity.

DETAILED DESCRIPTION:
The ketogenic diet has recently gained popularity as an effective dietary plan for weight management. Some of the cited benefits include a reduction in appetite and hunger, as well as improvements in fat oxidation leading to weight loss. Remarkably, some studies have also demonstrated increases in high-density lipoprotein (HDL) cholesterol and decreases in triglyceride levels, which point to a reduction in cardiovascular disease (CVD) risk.

In spite of these, there are still widespread concerns regarding the potentially high proportion of total and saturated fats derived from ketogenic diets owing to the high-fat and moderate-protein nature. These are associated with elevated low-density lipoprotein (LDL) cholesterol levels which may offset the purportedly lower CVD risk, especially in obese individuals. Furthermore, few randomised controlled trials (RCTs) have placed emphasis on the reduction of saturated fat, leading to confounding effects on the safety of the traditional ketogenic diet. To address the research gap, our study aims to assess the effect of a calorie-restricted healthy ketogenic diet, as compared to a calorie-restricted low fat diet on weight loss and metabolic outcomes among Asian individuals with obesity.

In this randomized controlled trial, participants will be randomly assigned to either the healthy ketogenic diet (HKD) or low fat calorie-restricted diet (LFD) using computer-generated random sequencing. Both the HKD and LFD groups will attend group workshops conducted by dietitians at weeks 1, 3, 5, 7, and thereafter at 6-week intervals over the course of a 6-month period.

The participants will be recommended to achieve their incremental daily step count goal from 3,000, 7,000 to 10,000 to promote increased physical activity, as per their tolerance. All participants are to provide for their own meals and follow a calorie-restricted diet with emphasis on the consumption of healthy fats and the reduction of saturated and trans fats in both diets.

Participants in the HKD group will be advised to follow a calorie-restricted healthy ketogenic diet (n=35), with a maximum of 50g net carbohydrate intake daily. Those in the control group will be instructed to follow a calorie-restricted low fat diet (LFD) (n=35). Calorie prescriptions for both diets were calculated based on the Schofield equation, adjusted with a deficit of 500 kcal daily to promote weight loss. Participants will also be recommended to use the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, steps count and to aid in their adherence to the diet and physical activity recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 27.5 to 40 kg/m2
* Aged 21 to 65 years

Exclusion Criteria:

* Individuals with type 1 diabetes or type 2 diabetes on insulin
* heart failure
* active cancer or in remission for less than 5 years
* advanced kidney disease
* hypothyroidism
* pregnancy
* depression
* untreated anemia, known thalassaemia, or other blood disorders.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | 6 months
  Weight changes post intervention

SECONDARY OUTCOMES:
Body weight | 3 months and 1 year
  Weight changes at follow up appointments
Blood pressure | 3 months, 6 months, 1 year
  Systolic and diastolic changes at follow up appointments
Hemoglobin A1c | 3 months, 6 months, 1 year
  HbA1c changes at follow up appointments
Fasting blood glucose | 3 months, 6 months, 1 year
  Fasting blood glucose changes at follow up appointments
Total cholesterol | 3 months, 6 months, 1 year
  Cholesterol changes at follow up appointments
Low-density lipoprotein cholesterol | 3 months, 6 months, 1 year
  Cholesterol changes at follow up appointments
High-density lipoprotein cholesterol | 3 months, 6 months, 1 year
  Cholesterol changes at follow up appointments
Triglycerides | 3 months, 6 months, 1 year
  Triglycerides changes at follow up appointments
Alanine transaminase | 3 months, 6 months, 1 year
  ALT changes at follow up appointments
Aspartate transaminase | 3 months, 6 months, 1 year
  AST changes at follow up appointments
Plasma 3-hydroxybutyrate (3-OHB) | 3 months, 6 months, 1 year
  Blood ketones at follow up appointments
Dietary intake | 3 months, 6 months, 1 year
  Nutrients intake by assessing 2-day food diaries
Physical activity | 3 months, 6 months, 1 year
  Physical activity frequency and intensity via self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Su Lin Lim, PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will remain confidential and only accessible via lock and keys by the researchers.